CLINICAL TRIAL: NCT03524404
Title: BRInging the Diabetes Prevention Program to GEriatric Populations(BRIDGE): a Pilot Study to Test the Usability and Effectiveness of a Telehealth Adaption of the Diabetes Prevention Program (DPP) in a Community of Older Adults
Brief Title: BRInging the Diabetes Prevention Program to GEriatric Populations - PILOT
Acronym: BRIDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-00229
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetes Prevention Program (DPP) (Experimental): Live stream the first six sessions of the Diabetes Prevention Program (DPP) curriculum to Senior Planet on a weekly basis, The webinars will be about 1 hour long, led by a certified DPP educator, and live-streamed to the senior center. Participants will have weekly weigh-ins and meet with a research assistant led focus group following two out of the six sessions to discuss program acceptability.
  Interventions: Behavioral: 6 Week Intervention

INTERVENTIONS:
Behavioral: 6 Week Intervention — Weekly interactive webinars based on the DPP curriculum at senior center.

SUMMARY:
The purpose of this pilot study is to test the feasibility of implementing a telehealth adaption of the Diabetes Prevention Program (DPP) intervention among 30 NYC senior center members. The intervention will be conducted through 6 weekly webinars with a certified DPP coach. Participants will receive a binder and physical activity tracker to complete self-monitoring of diet and physical activity. The primary outcome is feasibility and acceptability of the intervention measured by workshop attendance and focus group feedback. Secondary outcomes include changes in diet, physical activity, and weight.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥ 60 years
* Diabetes Risk Score >=5

Exclusion Criteria:

* Decisional incapacity to consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Program engagement | 8 Weeks
  calculated by subtracting attending study visits from those enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Beasley, MD, Principal Investigator — Jeannette.Beasley@nyumc.org
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Beasley JM, Kirshner L, Wylie-Rosett J, Sevick MA, DeLuca L, Chodosh J. BRInging the Diabetes prevention program to GEriatric populations (BRIDGE): a feasibility study. Pilot Feasibility Stud. 2019 Nov 11;5:129. doi: 10.1186/s40814-019-0513-7. eCollection 2019. PMID 31741744